CLINICAL TRIAL: NCT06373029
Title: Deep Learning-enabled Ultrasound Classification of Anterior Talofibular Ligament Injury in China: A Prospective, Multicentre, Diagnostic Study
Brief Title: Deep-learning Enabled Ultrasound Diagnosis of Anterior Talofibular Ligament Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Jiaan, Chairman, Peking University People's Hospital
Other Study IDs: 2023PHB211-001(2)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Ultrasound; Anterior Talofibular Ligament; Deep Learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — The investigators made ultrasound examinations to the participants to test whether the model could improve their diagnostic accuracy

SUMMARY:
Ultrasound (US) is a more cost-effective, accessible, and available imaging technique to assess anterior talofibular ligament (ATFL) injuries compared with magnetic resonance imaging (MRI). However, challenges in using this technique and increasing demand on qualified musculoskeletal (MSK) radiologists delay the diagnosis. The investigators have already developed a deep convolutional network (DCNN) model that automates detailed classification of ATFL injuries. The investigators hope to use the DCNN in real-world clinical setting to test its diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years old
* patients who underwent an acute ankle sprain
* patients with a surgery results of the sprained ankle

Exclusion Criteria:

* age< 18 years old
* patients with a previous history of ankle surgery
* patients with ankle tumors
* patients with a previous history of rheumatoid arthritis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As mentioned above
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
classification of ATFL injury | Baseline
  ultrasound classification of ATFL injury versus surgery results

CONTACTS AND LOCATIONS:
Overall Officials: Jiaan Zhu, Dr, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. Evidence review for the 2016 International Ankle Consortium consensus statement on the prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1496-1505. doi: 10.1136/bjsports-2016-096189. Epub 2016 Jun 3. PMID 27259753
- [Background] Kramer Z, Woo Lee Y, Sherrick R. Acute Ankle Sprains. Clin Podiatr Med Surg. 2023 Jan;40(1):117-138. doi: 10.1016/j.cpm.2022.07.008. PMID 36368838